CLINICAL TRIAL: NCT01610947
Title: Effect of Spacing of Anti-TNF Drugs in Ankylosing Spondylitis With Low Disease Activity: a Randomized Controlled Trial
Brief Title: Effect of Spacing of Anti-TNF Drugs in Ankylosing Spondylitis With Low Disease Activity
Acronym: SPACING
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 8785
Record Dates: First submitted 2012-05-24; First posted 2012-06-04 (Estimated); Last update posted 2021-10-19 (Actual); Status verified 2021-10

CONDITIONS: Spondyloarthritis
Keywords: Spondyloarthritis; Anti-TNF; Adalimumab; Etanercept; Infliximab
MeSH Terms: conditions — Spondylarthritis | interventions — Adalimumab; Etanercept; golimumab; Infliximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Maintain (Active Comparator): Continuation of usual treatment with fixed intervals according to standard recommendations
  Interventions: Drug: Adalimumab, Etanercept, Golimumab or infliximab
- Spacing (Active Comparator): Progressive spacing of injections according to disease activity observed during follow-up and predefined protocol.
  Interventions: Drug: Adalimumab, Etanercept, Golimumab or infliximab

INTERVENTIONS:
Drug: Adalimumab, Etanercept, Golimumab or infliximab — Continuation of usual treatment with fixed intervals according to standard recommendations
  Arms: Maintain
Drug: Adalimumab, Etanercept, Golimumab or infliximab — Progressive spacing of injections according to disease activity observed during follow-up and predefined protocol
  Arms: Spacing

SUMMARY:
Patients with spondyloarthritis, already treated by TNF blocker (adalimumab, etanercept or infliximab), and in stable low disease activity for at least 6 months, will be randomized into 2 groups: either keeping on their usual treatment with stable doses or progressive spacing of injections of their treatment. Follow-up will be done every 3 months during 12 months, with regular monitoring of disease activity and, in patients from the group "spacing", modification of the rhythm of injections according to health state and predefined protocol.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with spondyloarthritis according to ASAS criteria
* Stable low disease activity for at least 6 months
* Already treated by TNF blocking drug (adalimumab, etanercept or infliximab)

Exclusion Criteria:

* Raised acute phase reactants
* participation in another clinical trial
* Structural progression of peripheral joint damage
* Scheduled surgery within 12 months
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 398 (Actual)
Dates: Start 2012-05-14 (Actual); Primary Completion 2018-10-18 (Actual); Study Completion 2018-10-18 (Actual)

PRIMARY OUTCOMES:
Proportion of patients remaining in low disease activity | 12 months

SECONDARY OUTCOMES:
Medico-economic comparison of arms | 12 months
  The cost-efficacy ratio will be compared between the 2 arms (maintain and spacing). The objective is to see if the spacing of the treatments will allow a better tolerance and reduce the cost due to the treatments.To assess this cost-efficacy ratio, questionnaires will be used (quality of life SF36, medico-economic Euroqol).

CONTACTS AND LOCATIONS:
Locations (1):
- Lapeyronie Hospital, Montpellier, France